CLINICAL TRIAL: NCT06701006
Title: Integrated Screening and Safety Planning (ISSP) for Adolescents With Suicidal Thoughts
Brief Title: Integrated Suicide Supports and Safety Planning for Youth
Acronym: ISSP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Laura Richardson, Professor of Pediatrics, University of Washington
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00020199; P50MH129708 (NIH)
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Suicidal Ideation; Suicidal Behavior
Keywords: adolescents; young adults; suicide prevention; health services research
MeSH Terms: conditions — Suicidal Ideation; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: This trial will use a pre- post- sequential design in which each clinic has a control period (usual care), followed by provider training, and then an intervention period (usual care plus Jaspr app).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention)
- Integrated skills and safety planning app (Experimental): Use of Jaspr app in clinic + at home
  Interventions: Other: Integrated skills and safety planning app

INTERVENTIONS:
Other: Integrated skills and safety planning app — This is a digital app that includes supported safety planning resources in clinic as well as coping skills and lived experience videos for adolescents, young adults and parents/caregivers that can be accessed in clinic or at home.
  Other Names: Jaspr
  Arms: Integrated skills and safety planning app

SUMMARY:
The goal of this clinical trial is to evaluate an app to help keep teens and young adults with suicidal thoughts safe. The app includes a safety plan created by adolescents and healthcare providers in the clinic, and videos to encourage supportive communication and skills for teens and young adults to stay safe. The main question it aims to answer is whether the use of an app can increase youth suicide-related coping for youth with suicidal ideation, parent suicide prevention self-efficacy, and healthcare provider self-efficacy in suicide management. Researchers will compare usual care to usual care with the app. Participants, including adolescents, their caregivers and healthcare providers, will use the ISSP app (if assigned to that group) and complete three online surveys.

DETAILED DESCRIPTION:
The current study aims to evaluate the Jaspr app relative to usual care among youth (ages 13-21 years) who indicate suicidal ideation in pediatric outpatient medical settings. The Jaspr app includes supported safety planning between the young person and the healthcare provider, as well as skills and support videos for youth and caregivers intended to increase coping and decrease distress with an opportunity to access these resources through an at home app. Adolescents, parents, and clinicians will participate in the project to assess the effectiveness of Jaspr augmenting usual care, compared to usual care alone. The study will use a pre-post design in which each clinic begins with a control period and then transitions to the addition of Jaspr following healthcare provider training on use of the app. Participants and their parents will receive study assessments at baseline, 1-month, and 2-month follow up timepoints, and healthcare providers complete a survey at baseline, the end of the control period, and the end of the intervention period. Study assessments with youth will ask about coping, suicidal ideation and severity, anxiety and depression, service utilization, functional impairment, access to lethal means, and acceptability of the app. Study assessments for parents will ask about their self-efficacy in managing their youth's suicidality, acceptability of the app, and service utilization for the youth. Healthcare providers will complete surveys assessing their self-efficacy in managing youth suicidality. Youth, their legal guardian, and healthcare providers each assent/consent to participate in the research procedures.

ELIGIBILITY:
Youth Inclusion Criteria:

* Age 13 -21 years, an Ask Suicide Questions (ASQ) screen score of 1-5 with no current plan or intent requiring acute referral to higher level care and/or a risk level of suicidal thoughts and behaviors (STB) that constitutes the need for higher level assessment (such as the BSSA or C-SSRS) and/or a safety plan, as determined by an HCP because of a risk screener or a clinical interaction
* Parents/guardians: One "parent" per AYA will also be invited to participate.
* HCPs: All HCPs in participating clinics who may conduct assessments of SI (physicians, nurse practitioners/physician's assistants, social workers, nurses, psychologists) will be invited to participate.
* All subjects must have access to the internet and a computer or tablet device.

Youth Exclusion Criteria:

* Concurrently enrolled in an affiliated Suicide Care Research Center study, no phone access, or non-English speaking.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Youth Suicide-Related Coping | Baseline, 1 month, 2 month
  Total Score on the 17-item Youth Suicide-Related Coping Scale
Parent suicide prevention self-efficacy | Baseline, 1 month, 2 month
  Total score on the Parent suicide prevention self-efficacy scale
Healthcare provider self-efficacy in suicide management | Baseline, end of control period, and end of intervention period
  Total score on the Provider suicide Intervention Questionnaire

SECONDARY OUTCOMES:
Safety Plan Quality | Up to 1 month
  Safety Planning Scoring Algorithm (SPISA) based on youth medical chart review
Youth Suicide Severity | Baseline, 1 month, 2 month
  Total score on the online self-report version of the Columbia Suicide Severity Rating Scale (C-SSRS)
Youth Anxiety Symptoms | Baseline, 1 month, 2 month
  Total Score on Youth Self-Reported Generalized Anxiety Disorder -7 item scale
Intervention Acceptability | Baseline, 1 month, 2 month
  Youth and Parent Report on the Acceptability of Intervention Measure (AIM)
Functional Impairment | Baseline, 1 month, 2 month
  Total score on the youth reported EQ-5D-Y quality of life measure
Youth Suicidal ideation | Baseline, 1 month, 2 month
  Total Score on the Harkavy Asnis Suicide Scale ideation subscale (HASS-I),
Youth Depressive Symptoms | Baseline, 1 month, 2 month
  Total score on the Patient Health Questionnaire 9

OTHER OUTCOMES:
Access to Lethal Means | 1 month
  BRFSS Module 17 - Youth report of access to a firearm
Intervention Feasibility | Baseline, 1 month, 2 month
  Healthcare Provider Report on the Feasibility of Intervention Measure (FIM)
Mental Health Services Use | Baseline, 2 months
  Dichotomous rating of any mental health service use following baseline using chart review or indication based on parent or youth report on the Services Assessment for Children and Adolescents (SACA)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Richardson, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share required elements with the NIMH NDA.